CLINICAL TRIAL: NCT03868033
Title: Department of Orthopedics, National Taiwan University Hospital
Brief Title: Denosumab Sequential Therapy
Acronym: DST
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201811067MIPC
Record Dates: First submitted 2019-03-06; First posted 2019-03-08 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2023-09

CONDITIONS: Osteoporosis
Keywords: Osteoporosis; Denosumab; Zoledronate; Bone mineral density
MeSH Terms: conditions — Osteoporosis | interventions — Zoledronic Acid; Denosumab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Continuous Denosumab (Experimental): Continuous anti-resorptive therapy by Denosumab for 2 years
  Interventions: Drug: Denosumab
- Zoledronic acid to Denosumab (Experimental): treat with Zoledronic acid for one year and then shift to Denosumab for another one year
  Interventions: Drug: Zoledronic Acid; Drug: Denosumab
- Continuous Zoledronic acid (Experimental): Continuous anti-resorptive therapy by Zoledronic acid for 2 years
  Interventions: Drug: Zoledronic Acid
- Zoledronic acid to observation (Experimental): treat with Zoledronic acid for one year and then close follow up by bone turn over marker.
  resume another dose of Zoledronic acid if elevated CTX level above normal range
  Interventions: Drug: Zoledronic Acid

INTERVENTIONS:
Drug: Zoledronic Acid — Use Zoledronic acid as a sequential therapy after denosumab treatment for more than 2 years
  Other Names: Aclasta
  Arms: Continuous Zoledronic acid; Zoledronic acid to Denosumab; Zoledronic acid to observation
Drug: Denosumab — Continuous Denosumab treatment in arm 1 for two years or as a 2nd year treatment in arm 2 for one year
  Other Names: Prolia
  Arms: Continuous Denosumab; Zoledronic acid to Denosumab

SUMMARY:
Denosumab is a potent anti-resorptive agent and is now widely used in the treatment of osteoporosis. Although denosumab has excellent effect to increase bone mass and prevent fracture in FREEDOM study with very low complications, even up to ten years, it's effect is reversible. After holding the drug, circulating denosumab levels fall rapidly, and bone resorption reaching twice baseline levels for about 6 months. How to prevent bone loss after denosumab therapy is an important issue, especially when considering the compliance, persistence, or other comorbidities of the patient. We want to verify if zoledronic acid could be used as a sequential therapy after denosumab to prevent rapid bone loss by randomized clinical trial.

DETAILED DESCRIPTION:
Denosumab is a monoclonal antibody directed against the protein RANK-L, the principal regulator of osteoclast development. Thus, it acts as a potent anti-resorptive agent and is now widely used in the treatment of osteoporosis. Because it's easily to be used with very low risk of complications, patient has better compliance and persistence of denosumab than bisphosphonates. It's market share increasing very rapidly in Taiwan.

Although denosumab has excellent effect to increase bone mass and prevent fracture in FREEDOM study with very low complications, even up to ten years, it's effect is reversible. After holding the drug, circulating denosumab levels fall rapidly, and bone resorption reaching twice baseline levels for about 6 months. Over the first 12 months off therapy, all the bone density gained on treatment is lost4. According to previous meta-analysis study, although the persistence of denosumab therapy is better than bisphosphonates, only 62% patients keep the treatment after two years. We could image how low the persistence is after five-year or ten-year treatment in the real world.

How to prevent bone loss after denosumab therapy is an important issue, especially when considering the compliance, persistence, or other comorbidities of the patient. There is only one randomized controlled trial dealing with this problem, although the primary goal of the study is designed to compare the compliance and persistence1. After switching from denosumab to alendronate for one year, bone mineral density does not decrease rapidly, although there is mild elevation of bone turn over marker.

We want to verify if zoledronic acid could be used as a sequential therapy after denosumab to prevent rapid bone loss by randomized clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Postmenopausal women
2. Men >50-year-old
3. After Denosumab treatment ≥ 2 years due to osteoporosis

Exclusion Criteria:

1. Patientshadeverusedantiosteoporosismedications other than Dmab
2. Estimated glomerular filtration rate <35 ml/min.
3. Malignancy
4. Continuous steroid treatment, hormone therapy or other medical treatment affecting bone metabolism
5. Secondary osteoporosis
6. Metabolic bone diseases
7. Contraindications to ZOL
8. Patients older than 80 years old
9. Hypocalcemia

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2019-04-12 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Changes of lumbar spine, total hip and femoral neck bone mineral density | baseline, 1 year, 2 year
  Changes of lumbar spine, total hip and femoral neck bone mineral density from baseline

SECONDARY OUTCOMES:
Change of bone turnover marker | baseline, 6 months, 12 months, 15 months, 18 months, 24 months
  Changes of bone turnover marker, including C-terminal telopeptide of type I collagen (CTX) and propeptide of procollagen type I (P1NP)
Clinical osteoporotic fracture | baseline, 1 year, 2 year
  Incidence of clinical osteoporotic fracture

CONTACTS AND LOCATIONS:
Overall Officials: Shau-Huai Fu, doctor, Principal Investigator — Department of Orthopedics, National Taiwan University Hospital Yunlin Branch; Chia-Che Lee, Principal Investigator — Department of Orthopedics, National Taiwan University Hospital
Locations (1):
- Department of Orthopedics, National Taiwan University Hospital, Taipei, N/A = Not Applicable, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee CC, Wang CY, Yen HK, Hung CC, Lai CY, Hu MH, Wang TM, Li CY, Fu SH. Zoledronate Sequential Therapy After Denosumab Discontinuation to Prevent Bone Mineral Density Reduction: A Randomized Clinical Trial. JAMA Netw Open. 2024 Nov 4;7(11):e2443899. doi: 10.1001/jamanetworkopen.2024.43899. PMID 39527056
- [Derived] Lee CC, Wang CY, Hung CC, Huang CC, Li CY, Chen HY, Chang YL, Tseng WJ, Wang TM, Yang RS, Wong TH, Fu SH. A Multi-Institutional Randomized Controlled Trial to Investigate Whether Zoledronate Prevents Bone Loss After Discontinuation of Denosumab: The Study Protocol of Denosumab Sequential Therapy (DST) Trial. Front Med (Lausanne). 2021 Sep 8;8:717168. doi: 10.3389/fmed.2021.717168. eCollection 2021. PMID 34568375